CLINICAL TRIAL: NCT06068855
Title: BOTOX® (Botulinum Toxin Type A) for the Reduction of Masseter Muscle Prominence: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: A Study to Assess the Effectiveness of BOTOX (Botulinum Toxin Type A) Injections for the Change of Masseter Muscle Prominence in Adult Participants
Acronym: MMP EU P3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M23-123; 2022-500568-37-00 (Other: EU CT)
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Masseter Muscle Prominence
Keywords: Masseter Muscle Prominence; BOTOX; Botulinum Toxin Type A
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Double-Blind Period: Botox (Experimental): Participants will receive 6 intramuscular injections of BOTOX to the masseter on Day 1.
  Interventions: Drug: BOTOX
- Open-Label Period: Botox (Experimental): Participants who are eligible for retreatment will be given open-label BOTOX on Day 180 and will be followed for up to 6 months
  Interventions: Drug: BOTOX
- Double Blind Period: Placebo (Placebo Comparator): Participants will receive 6 intramuscular injections of Placebo to the masseter on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BOTOX — Intramuscular Injections
  Other Names: Botulinum Toxin Type A
  Arms: Double-Blind Period: Botox; Open-Label Period: Botox
Drug: Placebo — Intramuscular Injections
  Arms: Double Blind Period: Placebo

SUMMARY:
The masseter muscle is one of the muscles in the lower face used for chewing. Prominence of the masseter muscle can appear as a widened and square lower face shape, which is an aesthetic concern for individuals who prefer a narrower and more ovoid lower face shape. Treatments are available for masseter muscle prominice (MMP), but researchers are looking for new non-surgical treatments. This study will assess adverse events and effectiveness of BOTOX in adult participants with MMP.

BOTOX is being investigated for the treatment of MMP. Participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is 1 in 4 chance that participants will be assigned to placebo. Around 248 adult participants with MMP will be enrolled in the study at approximately 30 sites in Europe.

Participants will receive either BOTOX or Placebo administered as 6 intramuscular injections to the masseter on Day 1. Participants who are eligible for retreatment will be given BOTOX on Day 180 and will be followed for up to 6 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 30 kg/m^2 using the calculation: BMI = weight (kg)/height (m)^2, rounded to the nearest whole number.
* Participants meets the following criteria:

  * Bilateral Grade 4 or Grade 5 MMP (identical grades for left and right side of the face), as determined at screening and at the Day 1 visit by the investigator using the MMPS.
  * Bilateral Grade 4 or Grade 5 MMP (identical grades for left and right sides of the face), as determined at the Day 1 visit by the participant using the MMPS-P.
  * MMP grades, as assessed by investigator and participant, do not need to be identical but have to be a minimum of Grade 4 with bilateral symmetry at Day 1.
* Participants who responded "A lot" or "Extremely" bothered by the appearance of their MMP as measured by the Bother Impact Assessment for Masseter Muscle Prominence (BIA-MMP) and attain a total score of ≥ 15 on the Lower Facial Shape Questionnaire - Impact Assessment (LFSQ-IA), determined at the Day 1 visit.

Exclusion Criteria:

* Has current intraoral infection, including infection of the mouth or gums, or facial skin infection requiring medical treatment in the opinion of the investigator.
* Has weakness of the masseter, pterygoid, or temporalis muscles due to trauma, facial nerve injury, or other condition that could interfere with normal chewing and jaw clenching, as determined by the investigator.
* Excess lower facial fat, jowling, loose or lax skin in lower face, or parotid gland prominence that could interfere with MMPS or MMPS-P grading, as determined by the investigator.
* Has medical condition that may put the participant at increased medical risk with exposure to BOTOX, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function.
* History of dental or surgical procedure for lower facial shaping or masseter muscle reduction.
* History of any soft tissue fillers in the jawline.
* Has prior exposure to botulinum toxin of any serotype to any part of the body (not including masseter muscle) within the 3 months prior to Day 1.
* History of or current TMJD, or presence of signs/symptoms of possible TMJD in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Achievement of 2-grade or more improvement from baseline on the Masseter Muscle Prominence Scale (MMPS) as assessed by the Investigator | Day 90
  The investigator assessed the severity of the participant's MMP using the MMPS 5-point scale where: 1=minimal (best), 2=mild, 3=moderate, 4=marked, and 5=very marked (worst).
Achievement of 2-grade or more improvement from baseline on the Masseter Muscle Prominence Scale - Participant (MMPS-P) as assessed by the Participant | Day 90
  The participant assessed the severity of their MMP using the MMPS-P 5-point scale where: 1=not at all pronounced (best), 2=mildly pronounced, 3=moderately pronounced, 4=pronounced, and 5=very pronounced (worst).

SECONDARY OUTCOMES:
Response of "Very Satisfied" or "Satisfied" on the Lower Facial Shape Questionnaire - Treatment Satisfaction Assessment (LFSQ-TXSAT) | Day 90 to Day 180
  The LFSQ-TXSAT measures the participant's satisfaction with the effect of treatment on the appearance of their lower face where 2=Very satisfied, 1=Satisfied, 0=Neither satisfied nor dissatisfied, -1=Dissatisfied, -2=Very dissatisfied.
Response of "Not at all bothered" or "A little bothered" on the Bother Impact Assessment for Masseter Muscle Prominence (BIA-MMP) | Day 90 to Day 180
  The BIA-MMP is a single item evaluation of how bothered the participant is by the appearance of their lower face where 0=Not at all bothered, 1=A little bothered, 2=Somewhat bothered, 3=A lot bothered, 4=Extremely bothered.
Change from baseline in lower facial volume (cm^3) | Day 90
  Lower facial volume is calculated from standardized images
Change from baseline in lower facial width (mm) | Day 90
  Lower facial width is calculated from standardized images
Change from baseline in Lower Facial Shape Questionnaire - Impact Assessment (LFSQ-IA) summary score | Day 90 to Day 180
  The LFSQ-IA is a 6-item assessment that measures psychosocial impact of the appearance of the lower face where 0= Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit and 4=Extremely.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (27):
- Belgium (4):
  - Da Vinci Clinic /ID# 246731, Beerse, Antwerpen
  - Evolve Clinic /ID# 246729, Schilde, Antwerpen
  - Universitair Ziekenhuis Brussel /ID# 246311, Jette, Brussels Capital
  - Lightfalls Clinic /ID# 247335, Melle, Oost-Vlaanderen
- Bulgaria (3):
  - Dermavist - Group Practice for Specialized Medical Care for Skin Disease /ID# 247630, Plovdiv
  - Medical Center Derma Vita EOOD /ID# 247327, Sofia
  - Medical Centre Dermatology Dr. Denkova EOOD /ID# 246591, Sofia
- France (4):
  - Mediti /Id# 246875, Antibes
  - Cabinet Dermatologie et Esthetique /ID# 246871, Cannes
  - Cabinet médical /ID# 246873, Paris
  - Cabinet de Chirurgie Plastique et Esthétique /ID# 246872, Toulouse
- Germany (5):
  - Hautok and Hautok-cosmetics /ID# 246600, Munich, Bavaria
  - Studienzentrum Theatiner46 /ID# 246601, Munich, Bavaria
  - Hautzentrum Koeln /ID# 247502, Cologne, North Rhine-Westphalia
  - Privatpraxis Dr. Hilton & Partner /ID# 246602, Düsseldorf, North Rhine-Westphalia
  - Universitaet Hamburg /ID# 247503, Hamburg
- Italy (3):
  - Azienda Unita Sanitaria Locale Latina /ID# 246835, Latina
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 246836, Roma
  - CRC - Centro Ricerche Cliniche di Verona S.r.l. /ID# 246834, Verona
- Spain (4):
  - Gavín Dermatólogos /ID# 252120, Vigo, Pontevedra
  - Clinica Alejandria /ID# 247380, Valencia, Valencia
  - Grupo Pedro Jaen /ID# 246485, Madrid
  - Clinica Robega /ID# 252239, Madrid
- United Kingdom (4):
  - Waverley Medical Practice /ID# 246432, Coatbridge, North Lanarkshire
  - Dr Nestor's Medical Cosmetic Centre /ID# 246437, Edinburgh
  - Interface Aesthetics Training Limited /ID# 248115, London
  - MediZen /ID# 246431, Sutton Coldfield

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-123